CLINICAL TRIAL: NCT04199962
Title: Genomic Approaches for Predicting Severity of Organ Dysfunction and Outcomes in Sepsis: a Prospective Cohort Study in Adult Critically Ill Patients With Sepsis
Brief Title: Genomics in Infection and Sepsis to Predict Organ Dysfunction and Outcomes in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lowell Ling, Clinical Lecturer, Chinese University of Hong Kong
Other Study IDs: 2019.372
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Infection; Pneumonia
Keywords: sepsis; infection; pneumonia; organ dysfunction; critical illness
MeSH Terms: conditions — Sepsis; Infections; Pneumonia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — single-cell suspension and plasma DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pneumonia without sepsis: adult patients with community acquired pneumonia change in SOFA score <2 (other than respiratory component)
- pneumonia with sepsis: adult patients with community acquired pneumonia change in SOFA score greater or equal to 2 (other than respiratory component)

SUMMARY:
This is a prospective cohort study using gene expression to study patients with infection and sepsis from pneumonia.

DETAILED DESCRIPTION:
This is a prospective cohort study using single cell transcriptomic profiling and plasma DNA tissue mapping on patients with pneumonia with or without sepsis. The major application of the investigator's study would be the discovery of gene expressions in different leucocytes and plasma DNA associated with each type of organ dysfunction in sepsis. These include cardiovascular, respiratory, hepatic, renal, neurological and haematological dysfunction. This would help prediction, diagnosis and development of therapies to treat sepsis. Leucocyte single cell transcriptome and plasma DNA tissue mapping may addresses the limitations of current evidence in 3 ways: (1) differentiate patients with uncomplicated pneumonia versus pneumonia with associated sepsis, (2) correlation with types and severity of organ dysfunction and (3) identifying molecular phenotypes of sepsis.

ELIGIBILITY:
Inclusion Criteria:

All of the following:

* newly admitted adult patients (≥ 18 years old)
* suspected community acquired pneumonia (CAP)
* compatible history of either sputum or cough or fever or rigors within 1 week
* chest X-ray infiltrates

Exclusion Criteria:

Any of the following:

* chest symptoms not solely accounted by pneumonia (cardiac failure, non cardiogenic pulmonary oedema, suspected pulmonary embolism, suspected secondary acute respiratory distress syndrome)
* immunosuppression
* current malignancy
* blood samples for gene expression could not be taken within 24 hours of admission
* prisoner/cogni tive impairment
* blood transfusion within 1 month
* hospitalization within 1 month

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted with community acquired pneumonia to a tertiary hospital in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-11-11 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
blood single cell transcriptome in infection and sepsis | within 24 hours of hospital admission
  comparison of single cell transcriptome between patients with uncomplicated pneumonia and pneumonia with sepsis

SECONDARY OUTCOMES:
blood single cell transcriptome as marker of organ dysfunction | at time points 0, 24 and 72 hours
  association of single cell transcriptome with different types and severity of organ dysfunction
plasma DNA | at time points 0, 24 and 72 hours
  comparison of plasma DNA with different types and severity of organ dysfunction
blood single cell transcriptome as predictor of clinical outcome | at time points 0, 24 and 72 hours
  association of single cell transcriptome with mortality and morbidity outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided